CLINICAL TRIAL: NCT01455311
Title: Evaluation of Image-guided Brushing of Pancreatic Cyst Wall in the Diagnosis of Cystic Pancreatic Tumors
Brief Title: Evaluation of Image-guided Brushing of Pancreatic Cyst Wall in Diagnosis of Cystic Pancreatic Tumors
Status: Terminated | Type: Observational
Why Stopped: funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-15973
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Tumors
Keywords: cystic pancreatic tumors; cystic pancreatic lesions; gastrointestinal; GI; EUS-FNA; EchoBrush®; cytology brush; endoscopic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cataloguing the proteins that are expressed in pancreatic cyst fluid will provide preliminary data that will be used for identification of candidate biomarkers to predict malignant transformation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Pancreatic Tumor Specimens: Specimen collection via EUS Guided Fine Needle Aspiration EchoBrush Sampling
  Interventions: Procedure: EUS Guided Fine Needle Aspiration; Procedure: EUS Guided EchoBrush Sampling

INTERVENTIONS:
Procedure: EUS Guided Fine Needle Aspiration — EUS-guided fine needle aspiration of the cyst fluid
  Other Names: EUS-FNA
Procedure: EUS Guided EchoBrush Sampling — EUS-guided brushing of the cyst wall
  Other Names: EchoBrush®; Endoscopic Ultrasound Cytology Brush

SUMMARY:
The goal of this study is to compare a sample of the cyst taken by a standard method (fine needle aspiration) to the sample taken by a new method using a device called the EchoBrush to see which method is more accurate at diagnosing cancer. We will also look at proteins (also called biomarkers) in the samples to see if they predict whether or not the cyst is cancerous.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be offered the study and those who consent will undergo Endoscopic Ultrasound (EUS) evaluation. All patients who consent to the study will undergo Endoscopic Ultrasound guided fine needle aspiration (EUS-FNA) and EUS guided EchoBrush. All patients will receive the recommended standard antibiotic prophylaxis (Ciprofloxacin 400 mg IV given 30 minutes prior to EUS) that is used prior to EUS-FNA of cystic pancreatic lesions and a prescription for oral Ciprofloxacin for 5 days post procedure (standard of care).

Participants with pancreatic cysts that are >10 mm but under 25 mm: These patients will undergo standard EUS-FNA of cyst fluid. From the first 19 participants, 0.5cc of aspirated cyst fluid will be sent for Proteomic analysis and the rest for cytology. EUS guided EchoBrush of the cyst wall will not be performed in this group of patients.

Participants with pancreatic cysts that are > 25 mm will undergo EUS guided Echobrush sampling of the cyst wall at the same time they undergo EUS-FNA. This will be done using the standard technique that is described below.

EUS guided cyst wall brushing and residual fluid aspirated after lavage with 2 cc of sterile normal saline The tip of the Echobrush and the saline used to lavage the cyst will be placed in the same specimen jar (Specimen 2) based on the discussion with published experts on the EchoBrush technique. It should be noted that the pancreatic cyst will be punctured with the 19G FNA needle only once to obtain the specimens mentioned above. A single pass with EUS-FNA is the standard of care for pancreatic cysts and this study does not alter standard of care. It should be noted that the two groups represent two samples from the same patient and same cystic lesion. Therefore each patient will serve as their own internal control. All patients will be considered for surgical resection. Patients who do not undergo surgical resection will be followed up per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet clinical criteria to undergo an Endoscopic Ultrasound (EUS) with fine needle aspiration (FNA).
* Pancreatic cystic lesion with a minimum diameter of 10 mm noted on a previous cross-sectional imaging modality
* All races will be eligible

Exclusion Criteria:

* Coagulopathy defined as an prothrombin time (PT) > 13.5 seconds or partial thromboplastin time (PTT) > 35 seconds
* Thrombocytopenia defined as a platelet count < 50, 000
* Known pancreatic cancer
* Recent pancreatitis defined as an episode of pancreatitis within 4 weeks of study enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study design will be prospective, and will include 48 consecutive adult patients between the ages of 18 and 85 years, with pancreatic cystic tumors identified on crosssectional imaging and referred for EUS evaluation per the following inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rank The Diagnostic Accuracy of Specimen | 12 Months
  The difference in diagnostic accuracy between the cytological grade of dysplasia on aspirated cyst fluid cytology (Specimen/ Group 1) and Echo Brush cytology (Specimen/ Group 2) when compared to surgical histology (Specimen 3).
  Specifically, the cellularity (scored 0 to 3) of specimen 1 will be compared to specimen 2 using the two-sample proportion test. In addition, the Spearman's rank correlation will be used to calculate the correlation between cytological grade of dysplasia of specimen 1 to specimen 3, and the correlation between specimen 2 to specimen 3.

SECONDARY OUTCOMES:
Cataloging Proteins | 12 Months
  Cataloging proteins that are expressed in the cyst fluid collected from Pancreatic cystic tumors using Proteomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shivakumar Vignesh, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States